CLINICAL TRIAL: NCT00519558
Title: Investigation of the Efficacy and Safety of NN-220 for 24 Weeks in Adults With Growth Hormone Deficiency
Brief Title: Growth Hormone Deficiency in Adults (GHDA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GHLIQUID-1518; JapicCTI-R070007 (Registry Identifier: JAPIC)
Record Dates: First submitted 2007-08-20; First posted 2007-08-22 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Growth Hormone Disorder; Adult Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Human Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: somatropin

SUMMARY:
This trial is conducted in Japan. The aim of this trial is to demonstrate superiority of the effect of NN-220 compared with that of placebo as assessed by the change in percent in truncal fat (kg) from baseline to 24 weeks' treatment (end of treatment) in patients with Growth Hormone Deficiency in Adults (GHDA).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with diagnosed GHD
* If the subject has a history of treatment of treatment for a tumour of pituitary or peripheral site, two years or more must have passed since completion of surgery, radiotherapy or other treatment, and recurrence of the underlying disease to be excluded
* Appropriate replacement therapy has been administered for more than 24 weeks for the treatment of other pituitary hormone deficiencies

Exclusion Criteria:

* Subject with a history of acromegaly
* Subject with diabetes mellitus
* Subject suffering from malignancy
* Several medical conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2003-05-31 (Actual); Primary Completion 2005-01-24 (Actual); Study Completion 2005-01-24 (Actual)

PRIMARY OUTCOMES:
Percent change in truncal fat (kg) from baseline | at 24 weeks (end of treatment)

SECONDARY OUTCOMES:
Change in total body fat, total LBM, etc. from baseline to 24 weeks
Lipid-related laboratory tests (total cholesterol, HDL-cholesterol, LDL-cholesterol, and triglyceride)
IGF-I SDS, IGFBP-3 SDS, and IGF-I/IGFBP-3 molar ratio
Adverse events
Clinical laboratory tests
FPG, insulin, and HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Tokyo, Japan

REFERENCES:
- [Derived] Chihara K, Kato Y, Shimatsu A, Tanaka T, Kohno H. Efficacy and safety of individualized growth hormone treatment in adult Japanese patients with growth hormone deficiency. Growth Horm IGF Res. 2008 Oct;18(5):394-403. doi: 10.1016/j.ghir.2008.02.002. Epub 2008 Apr 18. PMID 18395480
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com